CLINICAL TRIAL: NCT03856164
Title: Use of Tranexamic Acid for Prevention of Hemorrhage in Cesarean Delivery
Brief Title: Tranexamic Acid for Prevention of Hemorrhage in Cesarean Delivery
Acronym: TXA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Olutoyosi Ogunkua, MD, Assistant Professor of Anesthesiology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU-2018-0315
Record Dates: First submitted 2019-02-21; First posted 2019-02-27 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Post Partum Hemorrhage; Fibrinolysis; Hemorrhage; Blood Loss
Keywords: Tranexamic acid; TXA; Anti-fibrinolytics; Postpartum hemorrhage; Obstetric hemorrhage; Fibrinolysis
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic acid (Active Comparator): Tranexamic Acid for intravenous administration.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Normal saline for intravenous administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Two doses of Tranexamic Acid (1 gram), diluted in 100 cc of normal saline. Administered intravenously at least 10 minutes prior to skin incision and repeated immediately after placental delivery.
  Other Names: Cyklokapron
  Arms: Tranexamic acid
Drug: Placebo — 100 mL of normal saline. Administered intravenously at least 10 minutes prior to skin incision and repeated immediately after placental delivery.
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
The investigators prepared a novel study of tranexamic acid (TXA) designed to estimate the quantity of blood loss in women undergoing elective repeat cesarean deliveries. This is the first trial to utilize a prophylactic dose of TXA prior to incision followed by a subsequent prophylactic dose at placental delivery in obstetric patients undergoing scheduled cesareans. The purpose of this study is to quantify blood loss during uncomplicated repeat cesarean deliveries with and without TXA. The central hypothesis is that TXA administration reduces blood loss and fibrinolysis in women undergoing repeat cesarean sections.

DETAILED DESCRIPTION:
Obstetric hemorrhage has been identified as a contributory cause for the United States' suboptimal and inequitable outcomes among pregnant women. As such, obstetric hemorrhage has become a formal focus point in a national agenda to improve maternal outcomes. Strategies to identify maternal hypovolemia and treating obstetric hemorrhage are undergoing organized scrutiny in many states including Texas. Tranexamic acid (TXA) treatment is receiving increased emphasis in obstetric care because TXA inhibits fibrinolysis. Increased clot stability offers the possibility of preventing blood loss (prophylaxis) as well as mitigating ongoing hemorrhage. TXA therapy has been principally studied in nonpregnant populations; results of studies in pregnant women have been lacking.

Tranexamic acid is an antifibrinolytic agent that acts as a competitive inhibitor at the lysine binding sites of plasminogen and inhibits the ability of protease plasmin to cleave the fibrin clot. In large randomized controlled trials, it has been reported to be effective in decreasing perioperative blood loss in a variety of circumstances primarily involving trauma patients. Shakur and co-authors in a trial of 20,000 non-pregnant trauma patients reported a significant reduction in all-cause mortality after TXA administration. In another large study (WOMAN Trial), 20,000 pregnant women with hemorrhage were randomized to TXA or placebo. TXA was associated with a significant decrease in death due to bleeding.

Tranexamic acid's role in treating hemorrhage have been widely studied in non-pregnant populations. Studies of TXA in obstetrics are limited. The American College of Obstetricians and Gynecologists believes the data is insufficient to recommend tranexamic acid for prophylaxis.

The investigators designed a randomized placebo-controlled trial comparing TXA dosing prior to incision for cesarean delivery with a repeat dose given at placental delivery. The purpose is to quantify blood loss during uncomplicated repeat cesarean deliveries with and without TXA. The investigators elected to study scheduled elective cesareans because such procedures are at low risk for profound hemorrhage. It is the intent to have a study cohort where the two treatment groups (TXA or placebo) are as comparable as possible, so the efficacy of TXA is not tested in women with highly variable volumes of obstetric hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Intrauterine pregnancy
2. Age ≥ 18
3. Gestation age ≥ 37 weeks 0 days
4. Scheduled cesarean delivery
5. Second or third cesarean delivery
6. Singleton pregnancy

Exclusion Criteria:

1. First cesarean delivery
2. Four or more cesarean deliveries
3. Intrauterine fetal death
4. Fetal anomalies
5. Documented coagulopathy (Elevated Prothrombin Time (PT), Elevated Partial Thromboplastin Time (PTT), Elevated International Normalized Ratio (INR))
6. Thrombocytopenia (Platelet count < 100k)
7. Internal bleeding, external bleeding, easy bruising
8. History of thrombotic event
9. Hypertension
10. Diagnosis of renal insufficiency (Creatinine> 1 mg/dL)
11. Insulin-treated diabetes
12. Suspected morbidly adherent placenta
13. Placenta previa
14. Multiple Gestations
15. BMI ≥ 50
16. Hematocrit ≤ 25
17. Blood transfusion within 24 hours prior to cesarean delivery
18. History of abnormal bleeding or blood disorder
19. Planned general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olutoyosi Ogunkua, M.D., Principal Investigator — UT Southwestern
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Society of Anesthesiologists Task Force on Perioperative Blood Management. Practice guidelines for perioperative blood management: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Blood Management*. Anesthesiology. 2015 Feb;122(2):241-75. doi: 10.1097/ALN.0000000000000463. No abstract available. PMID 25545654
- [Background] WHO Recommendations for the Prevention and Treatment of Postpartum Haemorrhage. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK131942/ PMID 23586122
- [Background] Carroli G, Cuesta C, Abalos E, Gulmezoglu AM. Epidemiology of postpartum haemorrhage: a systematic review. Best Pract Res Clin Obstet Gynaecol. 2008 Dec;22(6):999-1012. doi: 10.1016/j.bpobgyn.2008.08.004. Epub 2008 Sep 25. PMID 18819848
- [Background] GBD 2015 Maternal Mortality Collaborators. Global, regional, and national levels of maternal mortality, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1775-1812. doi: 10.1016/S0140-6736(16)31470-2. PMID 27733286
- [Background] WOMAN Trial Collaborators. Effect of early tranexamic acid administration on mortality, hysterectomy, and other morbidities in women with post-partum haemorrhage (WOMAN): an international, randomised, double-blind, placebo-controlled trial. Lancet. 2017 May 27;389(10084):2105-2116. doi: 10.1016/S0140-6736(17)30638-4. Epub 2017 Apr 26. PMID 28456509
- [Background] Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 183: Postpartum Hemorrhage. Obstet Gynecol. 2017 Oct;130(4):e168-e186. doi: 10.1097/AOG.0000000000002351. PMID 28937571
- [Background] Ducloy-Bouthors AS, Jeanpierre E, Saidi I, Baptiste AS, Simon E, Lannoy D, Duhamel A, Allorge D, Susen S, Hennart B. TRAnexamic acid in hemorrhagic CESarean section (TRACES) randomized placebo controlled dose-ranging pharmacobiological ancillary trial: study protocol for a randomized controlled trial. Trials. 2018 Mar 1;19(1):149. doi: 10.1186/s13063-017-2421-6. PMID 29490690
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Hernandez JS, Alexander JM, Sarode R, McIntire DD, Leveno KJ. Calculated blood loss in severe obstetric hemorrhage and its relation to body mass index. Am J Perinatol. 2012 Aug;29(7):557-60. doi: 10.1055/s-0032-1310528. Epub 2012 Apr 11. PMID 22495893
- [Background] Huissoud C, Carrabin N, Audibert F, Levrat A, Massignon D, Berland M, Rudigoz RC. Bedside assessment of fibrinogen level in postpartum haemorrhage by thrombelastometry. BJOG. 2009 Jul;116(8):1097-102. doi: 10.1111/j.1471-0528.2009.02187.x. Epub 2009 May 12. PMID 19459866
- [Background] Khan KS, Wojdyla D, Say L, Gulmezoglu AM, Van Look PF. WHO analysis of causes of maternal death: a systematic review. Lancet. 2006 Apr 1;367(9516):1066-1074. doi: 10.1016/S0140-6736(06)68397-9. PMID 16581405
- [Background] Main EK, Goffman D, Scavone BM, Low LK, Bingham D, Fontaine PL, Gorlin JB, Lagrew DC, Levy BS; National Partnership for Maternal Safety; Council on Patient Safety in Women's Health Care. National Partnership for Maternal Safety: Consensus Bundle on Obstetric Hemorrhage. Obstet Gynecol. 2015 Jul;126(1):155-62. doi: 10.1097/AOG.0000000000000869. PMID 26241269
- [Background] McCormack PL. Tranexamic acid: a review of its use in the treatment of hyperfibrinolysis. Drugs. 2012 Mar 26;72(5):585-617. doi: 10.2165/11209070-000000000-00000. PMID 22397329
- [Background] Molina RL, Pace LE. A Renewed Focus on Maternal Health in the United States. N Engl J Med. 2017 Nov 2;377(18):1705-1707. doi: 10.1056/NEJMp1709473. No abstract available. PMID 29091560
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] John M. Eisenberg Center for Clinical Decisions and Communications Science. Management of Postpartum Hemorrhage: Current State of the Evidence. 2016 Jul 12. In: Comparative Effectiveness Review Summary Guides for Clinicians [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2007-. Available from http://www.ncbi.nlm.nih.gov/books/NBK379234/ PMID 27512800
- [Background] Sentilhes L, Winer N, Azria E, Senat MV, Le Ray C, Vardon D, Perrotin F, Desbriere R, Fuchs F, Kayem G, Ducarme G, Doret-Dion M, Huissoud C, Bohec C, Deruelle P, Darsonval A, Chretien JM, Seco A, Daniel V, Deneux-Tharaux C; Groupe de Recherche en Obstetrique et Gynecologie. Tranexamic Acid for the Prevention of Blood Loss after Vaginal Delivery. N Engl J Med. 2018 Aug 23;379(8):731-742. doi: 10.1056/NEJMoa1800942. PMID 30134136
- [Derived] Ogunkua OT, Duryea EL, Nelson DB, Eddins MM, Klucsarits SE, McIntire DD, Leveno KJ. Tranexamic acid for prevention of hemorrhage in elective repeat cesarean delivery-a randomized study. Am J Obstet Gynecol MFM. 2022 Mar;4(2):100573. doi: 10.1016/j.ajogmf.2022.100573. Epub 2022 Jan 15. PMID 35038612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on admission for delivery at an academic center between June 2019 and January 2020. The first participant was enrolled on June 17, 2019, and the last participant was enrolled on January 10, 2020.
Pre-assignment Details: Of the 110 enrolled participants, all met inclusion criteria and were randomized.
Groups:
- Tranexamic Acid: Participants received two doses (1 gram) of tranexamic acid diluted in 100 mL of normal saline. Tranexamic acid was given intravenously at least 10 minutes prior to skin incision and repeated immediately after placental delivery.
- Placebo: Participants received 100 mL of normal saline. Administered intravenously at least 10 minutes prior to skin incision and repeated immediately after placental delivery.
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (5.2) | 28.7 (5.2) | 29.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 110
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black, non-Hispanic | 1 | 9 | 10
  White, non-Hispanic | 2 | 0 | 2
  Hispanic | 52 | 46 | 98
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110
Parity [Count of Participants; unit: Participants]
  Parity = 1 | 26 | 23 | 49
  Parity = 2 | 26 | 27 | 53
  Parity = 3 | 1 | 3 | 4
  Parity = 4 | 1 | 2 | 3
  Parity = 5 | 1 | 0 | 1
Body Mass Index (kg/m^2) [Count of Participants; unit: Participants]
  < 25 | 1 | 3 | 4
  25 - < 30 | 17 | 16 | 33
  30 - < 35 | 17 | 16 | 33
  35 - < 40 | 10 | 13 | 23
  > =40 | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Blood Volume Loss
Description: Total blood volume loss will be calculated in milliliters.
Time Frame: 24 hours postpartum.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 55 | 55
milliliters | 2274 (469) | 2407 (388)

2. Secondary Outcome: D-Dimer (µg/mL)
Description: Measured from blood sample collection.
Time Frame: Collection prior to first drug infusion, immediately before second infusion and 24 hours postpartum.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 55 | 55
µg/mL
  Before Surgery | 2.9 (1.5) | 4.0 (5.3)
  After Delivery | 2.4 (1.3) | 3.8 (4.7)
  P.O.D. 1 | 2.1 (1.2) | 4.3 (2.4)

3. Secondary Outcome: Fibrinogen (mg/dL)
Description: Measured from blood sample collection.
Time Frame: Collection prior to first drug infusion, immediately before second infusion and 24 hours postpartum.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 55 | 55
mg/dL
  Before Surgery | 563.5 (83.9) | 550.7 (68.2)
  After Delivery | 499.6 (77) | 484.9 (82.5)
  P.O.D. 1 | 527.4 (69.8) | 525.4 (86.1)

4. Secondary Outcome: Tissue Plasminogen Activator Antigen (ng/mL)
Description: Measured from blood sample collection.
Time Frame: Collection prior to first drug infusion, immediately before second infusion and 24 hours postpartum.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 55 | 55
ng/mL
  Before Surgery | 8.1 (3.6) | 8.2 (2.7)
  After Delivery | 9.0 (3.7) | 9.6 (2.9)
  P.O.D. 1 | 7.5 (3.7) | 7.4 (3.3)

5. Secondary Outcome: Plasminogen Activator Inhibitor-Type-1 (Units/mL)
Description: Measured from blood sample collection.
Time Frame: Collection prior to first drug infusion, immediately before second infusion and 24 hours postpartum.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 55 | 55
IU/mL
  Before Surgery | 81.8 (34.7) | 61.7 (33.8)
  After Delivery | 67.0 (32.3) | 63.3 (31.9)
  P.O.D. 1 | 20.7 (26.7) | 22.1 (28.5)

6. Secondary Outcome: Rotational Thromboelastometry INTEM and EXTEM Clotting Time
Description: Rotational thromboelastometry is a whole blood viscoelastic test that analyzes deficits in clotting factors, clot strength, and clot breakdown. EXTEM, INTEM, and FIBTEM tests measure the extrinsic pathway, intrinsic pathway, and fibrinogen levels, respectively. Compared to non-pregnant patients, FIBTEM/EXTEM/INTEM amplitudes and the FIBTEM maximum clot firmness are higher in pregnant women. The EXTEM and INTEM clotting time are shorter, indicating the relative hypercoagulability of pregnancy. Reference ranges for INTEM Clotting Time (100-240 seconds), INTEM Maximum Clot Firmness (50-72 millimeter), EXTEM Clotting Time (38-79 seconds), EXTEM Maximum Clot Firmness (50-72 millimeter), FIBTEM Maximum Clot Firmness (9-25 millimeter).
Time Frame: Collection prior to first drug infusion, immediately before second infusion and 24 hours postpartum.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 55 | 55
seconds
  Before Surgery INTEM Clotting Time | 149.7 (14.4) | 150.5 (14.2)
  After Delivery INTEM Clotting Time | 137.4 (18.3) | 140.7 (29.9)
  P.O.D. 1 INTEM Clotting Time | 145.1 (16.3) | 141.2 (16.4)
  Before Surgery EXTEM Clotting Time | 54.0 (5.1) | 56.1 (7.2)
  After Delivery EXTEM Clotting Time | 54.9 (6.3) | 56.3 (8.0)
  P.O.D. 1 EXTEM Clotting Time | 49.3 (5.3) | 50.2 (6.9)

7. Secondary Outcome: Rotational Thromboelastometry INTEM, EXTEM, FIBTEM Maximum Clot Firmness
Description: as for outcome 6
Time Frame: Collection prior to first drug infusion, immediately before second infusion and 24 hours postpartum.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 55 | 55
millimeter
  Before Surgery INTEM Maximum Clot Firmness | 69.3 (3.3) | 69.4 (3.7)
  After Delivery INTEM Maximum Clot Firmness | 68.9 (3.2) | 68.4 (5.5)
  P.O.D. 1 INTEM Maximum Clot Firmness | 68.8 (3.1) | 68.8 (3.8)
  Before Surgery EXTEM Maximum Clot Firmness | 70.8 (3.1) | 71.2 (3.5)
  After Delivery EXTEM Maximum Clot Firmness | 69.8 (3.1) | 69.6 (5.5)
  P.O.D. 1 EXTEM Maximum Clot Firmness | 70.5 (2.8) | 70.4 (4.0)
  Before Surgery FIBTEM Maximum Clot Firmness | 24.2 (3.8) | 23.9 (4.8)
  After Delivery FIBTEM Maximum Clot Firmness | 22.5 (4.1) | 22.0 (4.4)
  P.O.D. 1 FIBTEM Maximum Clot Firmness | 25.8 (4.7) | 25.0 (5.0)

ADVERSE EVENTS:
Time Frame: During patient admission, minimum of 3 days.
Description: Only serious adverse events were collected according to the study protocol
Arm/Group | Tranexamic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03856164/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03856164/SAP_001.pdf
  • Informed Consent Form (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03856164/ICF_002.pdf